CLINICAL TRIAL: NCT01651494
Title: A Phase 1 Clinical Study With Influenza Antiviral DAS181-F04: Double-Blind, Randomized, Placebo-Controlled, Multi Dose Study in Healthy Adults
Brief Title: Influenza Antiviral DAS-181-F04 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-0009; HHSN272201500007I
Record Dates: First submitted 2012-07-12; First posted 2012-07-27 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04-05

CONDITIONS: Influenza
Keywords: DAS181; Influenza; inhalation; inpatient clinic; Multi-Dose; recombinant neuraminidase
MeSH Terms: conditions — Influenza, Human; Respiratory Aspiration | interventions — oplunofusp

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DAS181-F04 (Active Comparator): DAS181-F04: 20 mg single-dose each day via inhalation for 3 days; 6 subjects
  Interventions: Drug: DAS181
- Placebo (Placebo Comparator): Placebo: 20 mg single-dose each day via inhalation for 3 days; 3 subjects
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DAS181 — DAS181-F04 is a recombinant neuraminidase that is delivered onto the cell surface of the upper and central airway topically and locally through an inhaler as an encapsulated dry powder. DAS181-F04; 20 mg single-dose each day via oral inhalation for 3 days; 6 subjects
  Arms: DAS181-F04
Other: Placebo — Placebo: White to off-white powder with Lactose Monohydrate and 5 % moisture; 20 mg single-dose each day via oral inhalation for 3 days; 3 subjects
  Arms: Placebo

SUMMARY:
This study will be a double-blind, randomized, placebo-controlled study of a single dose (20mg) of Influenza Antiviral DAS181-F04 for 3 days. The group of nine subjects will be randomly assigned to DAS181 or placebo at 2:1 ratios. Subjects will be admitted to the inpatient clinic at a minimum of the night prior to first dose. The subjects will stay in the inpatient clinic for the duration of dosing and one day after dosing, they will be required to come back for follow-up visits on study days 4, 6, 9, 16 (+/-1 day), 32 (+/-3 days), and 90 (+/-10 days). The safety parameters will include abnormal laboratory values, adverse events and clinical observations.

DETAILED DESCRIPTION:
This study will be a double-blind, randomized, placebo-controlled study. The subjects will receive a single-dose treatment of DAS181-F04 or placebo at a targeted delivered dose of 20mg each day for three days. The subjects will be evaluated on the day before the initial dose (Day -1) and randomly assigned to DAS181-F04 or placebo in a 2:1 ratio. Subjects will be evaluated prior to dosing on Days 0, 1 and 2. Additional follow-up evaluations will occur one day after completion of dosing (Day 3) and on Days 4, 6, 9, 16 (+/-1 day), 32 (+/-3 days) and 90 (+/-10 days). The primary objective is to determine the safety and tolerability of DAS181-F04 encapsulated dry powder compared to placebo when administered by oral inhalation using a dry powder inhaler (DPI) in healthy adults. The secondary objective is to investigate the pharmacokinetic and immunologic profile of DAS181 encapsulated dry powder dose to dose and compared to placebo when administered by oral inhalation using a DPI in healthy adults. A total of 9 subjects, healthy male and female subjects, ages 18 to 45 years will be enrolled. Subjects will be randomized 2:1 ratio, wherein 6 subjects will receive the active drug and 3 subjects will receive placebo. Subjects may be replaced if a subject withdraws within 7 days (Day 9) after receipt of the final study drug dose.

ELIGIBILITY:
Inclusion Criteria:

-Male and female subjects in good health in the opinion of the site Principal Investigator (PI) or sub-investigator as determined by vital signs, medical history, and a physical exam. -Subjects must be able to verbalize understanding of the consent form, provide written informed consent and verbalize willingness to complete study procedures. -Be 18 to 45 years of age (inclusive), at the time of screening. -Subjects must have a Body Mass Index (BMI) of 17.5-35. Actual lower weight limit may be 50 kg, if BMI is in the range indicated. -No history of smoking in the past six months, regardless of clinical relevance. -Electrocardiogram (ECG) with no clinically significant abnormalities recorded at screening visit: PR interval within 120 and 200ms, QRS interval < 120ms, and confirmed QTc interval </= 440ms. -Blood pressure within normal limits (systolic 86 - 140mmHg; diastolic 50 - 90 mmHg) and heart rate between 45 and 100 beats per minute. -Chest X-ray shows no clinically significant abnormalities. -Forced expiratory volume in 1 second (FEV1) will be greater than 80% predicted; note: only one baseline value for FEV1 can be used to support inclusion criterion. -Negative Human Immunodeficiency Virus (HIV), HBSAg, and Hepatitis C Virus (HCV) antibody screening tests. -Negative screening tests for: marijuana, cocaine metabolite, amphetamines, opiates, PCP, barbiturates, benzodiazepines, and ethanol. -Subjects with the following laboratory criteria within provided range (see Appendix B): --Hemoglobin --White blood cell (WBC) and platelet count --Alkaline phosphatase (ALKP), total bilirubin, alanine aminotransferase (ALT), --Serum glucose; note: if a non-fasting glucose is performed and is abnormal, a fasting glucose measurement may be obtained in its place; if this is within the provided range, then subject may be enrolled. --Serum creatinine --Activated partial thromboplastin time (APTT) and fibrinogen -Urine glucose and blood tested by dipstick urinalysis are negative. Urine protein tested by dipstick is negative or trace. Menstruating females failing inclusion due to positive urine dipstick blood may be retested following cessation of menses. -Female subjects must be post-menopausal (one year or greater without menses), surgically incapable of childbearing, or agreeable to practicing abstinence or utilizing two effective methods of birth control during the study period and for 12 weeks after study product administration. Acceptable methods may include: --Intrauterine device --Spermicide --Barrier contraception --Hormonal contraception -A female subject must have had a negative serum pregnancy test during the screening visit and a negative urine pregnancy test within 24 hours of drug dosing. -If male, agrees to use medically accepted form of contraception from time of enrollment to 12 weeks after study product administration. -Agrees not to drink alcohol or participate in strenuous physical activity or exercise from 24 hours prior to Day -1 through the Day 6 follow-up visit.

Exclusion Criteria:

-Have received any investigational drug or vaccine within 30 days prior to study drug dosing or have had a serious adverse reaction or hypersensitivity to any drug. -Is planning to participate in another clinical trial within 30 days after the last dose of DAS181. -Have received blood products within 6 months of study enrollment. -Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements. -Have been on a liquid protein diet in the last month. -Are allergic to lactose. -Have sickle cell disease. -Have used any prescription or nonprescription drugs, excluding hormonal contraception, within 7 days prior to admission unless approved by the site PI or sub-investigator. Subjects must be willing to refrain from taking non-study medication and herbal supplements during the study through Day 32 except those approved by the site PI or sub-investigator. -Existence of any surgical, medical or laboratory condition that, in the judgment of the site PI or sub-investigator, might interfere with the safety, distribution, metabolism, or excretion of the drug. -Subjects with current or a previous history of respiratory diseases (e.g., asthma, allergic rhinitis, chronic obstructive pulmonary disease (COPD), cystic fibrosis, emphysema, or anaphylaxis) requiring acute or chronic medication, as determined by the investigator through medical history evaluation and physical examination. -Subjects who have experienced a previous episode of acute upper respiratory tract infection, pneumonia, otitis, bronchitis, or sinusitis within 2 weeks prior to screening. -Subjects with concurrent sustained respiratory symptoms (runny nose, sore throat, sneezing, coughing, or wheezing). -Subjects who have an oral temperature above 37.8 degrees C (100 degrees F). -Subjects with cancer or history of hematologic malignancy. Cancer is defined as any active neoplastic disease, excluding noninvasive basal cell carcinoma. -Subjects who have a planned hospital admission for any cause and/or a planned surgical procedure within 30 days of initiation of the study. -Female subjects who are pregnant or breast-feeding. -Subjects who have donated or lost more than 500mL of blood in the three months prior to screening or who plan to donate blood during study participation. -Subjects who have clinically significant medical or psychological conditions that would compromise the subject's safety, influence the results of the study, affect the subject's ability to participate in the study, or impair the subject's ability to provide informed consent. -Subjects who have a history of drug dependence, or psychiatric illness within 2 years of study enrollment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2011-08-12 (Actual); Primary Completion 2012-09-18 (Actual); Study Completion 2012-09-18 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of multiple dose DAS181-F04 treatment (measured in adverse events, hematology, clinical chemistry, blood coagulation, haptoglobin, urinalysis, throat swab for bacterial culture, ECG, chest X-ray, and spirometric lung function) | up to day 90

SECONDARY OUTCOMES:
Immunogenicity responses: Blood samples for the immunogenetic profile of DAS181- F04 will be collected | Day 0, 32, and 90
Pharmacokinetic profile of DAS181- F04: Cmax, Tmax, Area under the curve (AUC (0-t)), t1/2, AUC (0-infinity), plasma clearance (CL) | Day 0-4, 6, 9, and 16

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Bayview Medical Center - Infectious Diseases, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Zenilman JM, Fuchs EJ, Hendrix CW, Radebaugh C, Jurao R, Nayak SU, Hamilton RG, McLeod Griffiss J. Phase 1 clinical trials of DAS181, an inhaled sialidase, in healthy adults. Antiviral Res. 2015 Nov;123:114-9. doi: 10.1016/j.antiviral.2015.09.008. Epub 2015 Sep 25. PMID 26391974